CLINICAL TRIAL: NCT07305441
Title: Impact Assessment of the Jockey Club REACH & Map Program for Hard-to-reach Older Adults in the Community: A Target Trial Emulation
Brief Title: Impact Assessment of the Jockey Club REACH & Map Program for Hard-to-reach Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REACH & MAP
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hard-to-Reach Elderly
Keywords: Hard-to-Reach, elderly, functional status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment status (Experimental): To account for time bias, each subject will be created with two clones at time zero and assigned each of the two clones to either treatment or no-treatment status, respectively. The treatment status in each evaluative endpoint (i.e., 1-month, 4-month, 10-month, and 13-month) is defined as subjects who have received the mapped intervention for the respective length of time since the time zero during which the intervention has just commenced.
  Interventions: Behavioral: Mapped intervention based on health status
- No-treatment status (No Intervention): To account for immortal time bias, each subject will be created with two clones at time zero and assigned each of the two clones to either treatment or no-treatment status, respectively. The corresponding no-treatment status is defined as subjects who have not received any mapped intervention for the corresponding length of time.

INTERVENTIONS:
Behavioral: Mapped intervention based on health status — Intervention will be conducted to improve lifestyle based on their needs which include 1) Home modification, 2) Lifestyle-based health promotion, 3) Geriatric symptom management, 4) Health counseling for chronic disease management, 5) Counseling-based service, 6) Social network optimization, 7) Social support optimization
  Arms: Treatment status

SUMMARY:
The goal of this study is to evaluate the impact of the Reach-and-Map project on increasing functional capacity to optimize the functional ability of the vulnerable group of "Hard-to-Reach" older adults through increase the compatibility between their intrinsic capacity and environment.

DETAILED DESCRIPTION:
The overall aim of this project is to conduct a comprehensive impact assessment of the Jockey Club (JC) Reach & Map Program, utilizing a framework based on the World Health Organization (WHO) Health Impact Assessment. The study will evaluate how the program influences health outcomes among hard-to-reach older adults by assessing changes in key health determinants. The findings will be disseminated to relevant stakeholders to inform future policy setting and service planning, and long-term monitoring will be undertaken to evaluate the extent to which the impact assessment influences decision-making in aged care service development.

The primary focus of the evaluation is on the functional abilities of older adults, including physical, cognitive, psychological, and social functioning. The assessment will also cover core outcomes such as quality of life, frailty, and health service use, alongside person-centered measures like loneliness and mental health. Given the diverse services received by beneficiaries, the study will account for structural and social health determinants-such as age, gender, socio-economic status, and chronic disease burden-as covariates in the analysis. In addition, the project will explore the broader effects of the JC Reach & Map Program on aged care service utilization and document both the experiences of service recipients and stakeholders involved.

Specifically, the study objectives are: (1) to evaluate the impact of the JC Reach & Map Program on frailty, quality of life, and health service use among hard-to-reach older adults, focusing on physical, cognitive, psychological, and social functions; (2) to explore the engagement experiences and perceptions of older adults regarding the services received, and their impact on well-being, community engagement, and social integration; and (3) to explore the experiences of service stakeholders in reaching and working with this population, as well as to gather their insights on ideal service models and policies for hard-to-reach older adults.

ELIGIBILITY:
Inclusion Criteria:

* age > 60
* able to participate in the impact assessment as evidence by a test score of > 6 on the Abbreviated Mental Test
* has the functional ability to engage in the digital intervention
* able to communicate with the researcher

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5500 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
EuroQoL-5 Dimension-5 Level | Changes from baseline to 1 month, 4 month, 10 month, and 13 month post-intervention.
  Measuring Health-related quality of life (HRQL) (range from -0.59 to 1.0), higher score indicates better quality of life
Short Physical Performance Battery | Changes from baseline to 1 month, 4 month, 10 month, and 13 month post-intervention.
  Measuring by (range from 0 to 12), with higher score indicating better physical performance
5-minute Montreal Cognitive Assessment (MoCA) | Changes from baseline to 1 month, 4 month, 10 month, and 13 month post-intervention.
  Measuring Cognitive function (range from 0 to 30), A score of 26 or over is considered to be normal.
7-item Memory Complaint Scale (MCS) | Changes from baseline to 1 month, 4 month, 10 month, and 13 month post-intervention.
  Measuring Subjective Memory Score (range from 0 to 14), lower score indicates better memory performance. No MCs (0-2), Mild MCs (3-6), Moderate MCs (7-10), Severe MCs (11-14).
3-item University of California, Los Angeles (UCLA) Loneliness Scale | Changes from baseline to 1 month, 4 month, 10 month, and 13 month post-intervention.
  Measuring Loneliness (range 3-9), higher score indicates greater loneliness.
The 8-item Geriatric Depression Scale | Changes from baseline to 1 month, 4 month, 10 month, and 13 month post-intervention.
  Measuring Depression (range 0 to 8), with higher score indicating higher risk of depression
8-item Social Connectedness Scale Revised | Changes from baseline to 1 month, 4 month, 10 month, and 13 month post-intervention.
  Measuring Social connectedness (range 0 to 48), <22 indicates lack of social connectedness

SECONDARY OUTCOMES:
Health service utilization | Changes from baseline to 1 month, 4 month, 10 month, and 13 month post-intervention.
  Self-developed checklist on community care service for older adults in Hong Kong
Health service utilization | From baseline to 1 month, 4 month, 10 month, and 13 month post-intervention.
  Self-developed checklist on health service utilization (including visit to out-patient clinic, emergency medical service, an in-hospital service in private and/or public sectors).
  [generic] With the consent from the participants, the above information will be retrieved from the electronic health record. Otherwise, self-report method will be used for collecting the data.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers.